CLINICAL TRIAL: NCT05365074
Title: Perioperative Outcomes in Patients Received Spinal Chloroprocaine for Hip or Knee Arthroplasty
Brief Title: Intrathecal Chloroprocaine for Lower Limb Arthroplasty
Status: Completed | Type: Observational
Sponsor: Hôpital de la Croix-Rousse (Other)
Collaborators: Hospices Civils de Lyon (Other)
Responsible Party: Principal Investigator, Mikhail Dziadzko, MD, PhD, Senior physician, Hôpital de la Croix-Rousse
Other Study IDs: CSE-HCL 22_729
Record Dates: First submitted 2022-04-18; First posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Lower Limb Arthroplasty Under Chloroprocaine Spinal Anesthesia
Keywords: chloroprocaine; total hip arthroplasty; total knee arthroplasty; unicompartmental knee arthroplasty; spinal anesthesia
MeSH Terms: interventions — chloroprocaine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- chloroprocaine anesthesia for arthroplasty: patients having predicted uncomplicated surgery for total or unicompartment knee arthroplasty of anterior access total hip arthroplasty, operated under spinal anesthesia with 50 mg of chloroprocaine
  Interventions: Drug: Chloroprocaine Injection

INTERVENTIONS:
Drug: Chloroprocaine Injection — Spinal anesthesia with 50 mg of 1% Chloroprocaine

SUMMARY:
This study evaluates the perioperative course in adult patients undergoing total or partial knee arthroplasty, or total hip arthroplasty under chloroprocaine spinal anesthesia.

DETAILED DESCRIPTION:
This study evaluates the failure rate of spinal anesthesia, the duration of surgical anesthesia, the needs for complementary intraoperative analgesia, the time for recovery, the incidence of urinary retention, postoperative nausea and vomiting, and length of stay in the recovery room in patients operated for knee or hip arthroplasty under spinal anesthesia with chloroprocaine 50 mg.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* with spinal anesthesia using 50 mg of chloroprocaine
* operated for total knee, unicompartment knee or anterior access hip arthroplasty
* in the period of years 2020 - 2021

Exclusion Criteria:

* expressed disagreement to to participate after receiving information notice

Age Groups: Child, Adult, Older Adult
Study Population: Adult patients operated for total knee, unicompartment knee or anterior access hip arthroplasty under chloroprocaine spinal anesthesia in the period of years 2020 - 2021
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
Spinal anesthesia failure | Day 0
  proportion of patients with the necessity to convert initially planned spinal anesthesia into general anesthesia

SECONDARY OUTCOMES:
Hemodynamic instability | Day 0
  proportion of patients with >20% changes in blood pressure and ou heart rate comparing to baseline
Need for sedation | Day 0
  proportion of patients requiring intraoperative sedation for uncomfortable conditions
Surgical block duration | Day 0
  time of regression of sensitive and motor spinal block
PACU analgesia requirement | Day 0
  morphine equivalent requirement in PACU for the postoperative pain
Urinary retention | 24 hours
  proportion of patients requiring urinary catheter
Postoperative nausea and vomiting | 24 hours
  proportion of patients having nausea and vomiting
Length of stay in recovery room | Day 0
  Length of stay in recovery room

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital de la Croix Rousse - Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No
IPD are protected by the French regulation and will not be shared